CLINICAL TRIAL: NCT05095194
Title: Influence of Capsular Tension Ring on IOL-capsular Complex After Cataract Surgery in Patients With High Myopia: a Clinical Observation Based on SS-OCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Yune Zhao, Vice president of Eye Hospital of Wenzhou Medical University, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20210929CTR
Record Dates: First submitted 2021-09-30; First posted 2021-10-27 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: High Myopia; Capsular Tension Ring
MeSH Terms: interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High myopia patients who had cataract surgery with IOL and capsular tension ring implantation (Experimental): The patients' axial length is over 26 mm and are diagnosed age related cataract The patients' age are over 50
  Interventions: Procedure: Cataract surgery with IOL implantation and with/without capsular tension ring implatation
- High myopia patients who had cataract surgery with IOL implantation (Experimental): The patients' axial length is over 26 mm and are diagnosed age related cataract The patients' age are over 50
  Interventions: Procedure: Cataract surgery with IOL implantation and with/without capsular tension ring implatation

INTERVENTIONS:
Procedure: Cataract surgery with IOL implantation and with/without capsular tension ring implatation — Patients in this study will receive cataract surgery with IOL implantation and capsular tension ring implantation or cataract surgery with IOL implantation

SUMMARY:
The IOL-capsular complex is formed after cataract surgery and intraocular lens (IOL) implantation.Early postoperative mechanical wrapping of the anterior and posterior capsules plays a significant role in preventing IOL decentration and tilt, as well as formation of the IOL-capsular complex which reduces the incidence of posterior cataract opacity. Capsular tension rings were first introduced in the early 1990s for loosening and tightening the lens bag and maintaining the equatorial contour of the bag after cataract surgery.Today, capsular tension rings of many different designs are in use.The capsular tension rings can be used in eyes with fragile and split zonular fibers, as well as pseudoexfoliation, high myopia, Marfan syndrome, mature cataract and lens subluxation.The capsular tension ring reduces the incidence of decentration and tilt of the IOL by reducing capsular contraction. In addition, multi-focus IOL implantation combine with capsular tension ring result in smaller high-order aberrations in our eyes compared to cataract surgery with multi-focus IOL implantation alone.For patients with high myopia, they often have a longer axial length and a larger capsule diameter, which reduces the rotational stability of the IOL and may lead to tilt ,decentration and displacement of IOL.Currently, there is no literature guidance to compare the results of cataract surgery combined with or without capsular tension ring implantation in patients with high myopia.Our hospital has Swept-source Optical Coherence Tomography ( SS-OCT,Casia2, TOMEY, Japan), which can accurately photograph the process of IOL capsule bending and the changes of lens position after cataract surgery. SS-OCT can be used to evaluate the influence of capsular tension ring on the dynamic changes of IOL-capsular complex in patients with high myopia after cataract surgery.

DETAILED DESCRIPTION:
The IOL-capsular complex is formed after cataract surgery and intraocular lens (IOL) implantation.Early postoperative mechanical wrapping of the anterior and posterior capsules plays a significant role in preventing IOL decentration and tilt, as well as formation of the IOL-capsular complex which reduces the incidence of posterior cataract opacity. Capsular tension rings were first introduced in the early 1990s for loosening and tightening the lens bag and maintaining the equatorial contour of the bag after cataract surgery.Today, capsular tension rings of many different designs are in use.The capsular tension rings can be used in eyes with fragile and split zonular fibers, as well as pseudoexfoliation, high myopia, Marfan syndrome, mature cataract and lens subluxation.The capsular tension ring reduces the incidence of decentration and tilt of the IOL by reducing capsular contraction. In addition, multi-focus IOL implantation combine with capsular tension ring result in smaller high-order aberrations in our eyes compared to cataract surgery with multi-focus IOL implantation alone.For patients with high myopia, they often have a longer axial length and a larger capsule diameter, which reduces the rotational stability of the IOL and may lead to tilt ,decentration and displacement of IOL.Currently, there is no literature guidance to compare the results of cataract surgery combined with or without capsular tension ring implantation in patients with high myopia.Our hospital has Swept-source Optical Coherence Tomography ( SS-OCT,Casia2, TOMEY, Japan), which can accurately photograph the process of IOL capsule bending and the changes of lens position after cataract surgery. SS-OCT can be used to evaluate the influence of capsular tension ring on the dynamic changes of IOL-capsular complex in patients with high myopia after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* The patients are diagnosed age related cataract with axial length over 26mm
* The patients' age over 50 years old
* The patients plan to receive cataract surgery in Eye hospital of Wenzhou Medical University
* The dialated pupils are over 6mm
* Patients are willing and able to complete the follow-ups.

Exclusion Criteria:

* Patients with other type of cataract
* Patients have complications in the surgery and after surgery
* Patients have other severe diseases of eyes

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
The position of IOL | The 1st day after surgery
  Evaluation of the position of IOL through tilt,decentration and the process of capsule bending.
The position of IOL | The 1st week after surgery
  Evaluation of the position of IOL through tilt,decentration and the process of capsule bending.
The position of IOL | The 1st month after surgery
  Evaluation of the position of IOL through tilt,decentration and the process of capsule bending.
The position of IOL | The 3rd month after surgery
  Evaluation of the position of IOL through tilt,decentration and the process of capsule bending.

CONTACTS AND LOCATIONS:
Locations (1):
- Eye Hospital of Wenzhou Medical College, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided